CLINICAL TRIAL: NCT01860703
Title: A Double-Blind, Randomized, Crossover, Thorough QT/QTc Trial to Evaluate the Potential of Deferiprone to Prolong the QT Interval in Healthy Subjects
Brief Title: Evaluation of Whether Deferiprone Affects QT Interval in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LA37-1111
Record Dates: First submitted 2013-05-06; First posted 2013-05-23 (Estimated); Results first posted 2014-11-12 (Estimated); Last update posted 2014-11-12 (Estimated); Status verified 2014-11

CONDITIONS: Prolonged QTc Interval
Keywords: Ferriprox®; LI; DFP; Deferiprone; Healthy Volunteers
MeSH Terms: interventions — Deferiprone; Long Interspersed Nucleotide Elements; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A - Maximum Therapeutic Dose (Experimental): Single dose of 33 mg/kg rounded to the nearest 250 mg of deferiprone tablets
  Interventions: Drug: Deferiprone
- Treatment Arm B - Supratherapeutic Dose (Experimental): Single dose of 50 mg/kg rounded to the nearest 250 mg of deferiprone tablets
  Interventions: Drug: Deferiprone
- Arm C - Placebo Control (Experimental): Single dose of matching deferiprone and moxifloxacin placebo tablets.
  Interventions: Drug: deferiprone matching placebo tablets; Drug: placebo
- Arm D - Positive Control (Experimental): Single dose of one 400 mg moxifloxacin tablet.
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: Deferiprone — Ferriprox 500 mg tablets
  Other Names: Ferriprox; L1
  Arms: Arm A - Maximum Therapeutic Dose; Treatment Arm B - Supratherapeutic Dose
Drug: deferiprone matching placebo tablets — deferiprone matching placebo tablets
  Other Names: Placebo
  Arms: Arm C - Placebo Control
Drug: moxifloxacin — Active control
  Other Names: Avelox
  Arms: Arm D - Positive Control
Drug: placebo — moxifloxacin-matching placebo
  Arms: Arm C - Placebo Control

SUMMARY:
Randomized, single-dose, double-blind, placebo and active controlled, four-period crossover study to evaluate the effect of deferiprone on QTc prolongation after administration of a single therapeutic (33 mg/kg) and supratherapeutic(50 mg/kg) oral doses of deferiprone in healthy volunteers as compared to placebo treatment.

DETAILED DESCRIPTION:
Post-marketing study to evaluate the effect of deferiprone and deferiprone 3-O-glucuronide on QTc prolongation in healthy volunteers after administration of a single therapeutic (33 mg/kg) and supratherapeutic (50 mg/kg) oral dose of deferiprone and moxifloxacin (Avelox®).

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy adult males or females, 18 - 45 years of age (inclusive).
2. Body weight ≥ 50 kg.
3. Body mass index (BMI) ≥ 19 and ≤ 32 kg/m2.
4. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical history, vital signs, physical examination).
5. Absolute neutrophil count (ANC) of >1.5x109/L.
6. 12-lead ECGs which have no clinically significant findings as judged by the Principal Investigator (PI) or the PI's designee at screening and check-in of each study period,including:

   1. Normal sinus rhythm (heart rate between 45 and 100 bpm);
   2. QTcF interval ≤ 450 msec;
   3. QRS interval ≤ 110 msec; and
   4. PR interval ≤ 220 msec.
7. Subject must be capable of providing written informed consent, and must voluntarily consent to participate in the study.
8. Willing to answer inclusion and exclusion criteria questionnaire at check-in.

Main Exclusion Criteria:

1. History or presence of significant respiratory, cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic,neurologic, or psychiatric disease.
2. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the PK of the investigational medicinal products (e.g. cholecystectomy, resections of the small or large intestine, febrile conditions, chronic diarrhea, chronic vomiting, endocrine disease, severe infections,acute inflammations, etc.).
3. Presence of liver impairment: aspartate aminotransferase (AST), alanine aminotransferase (ALT) above the normal reference range.
4. Presence of significant kidney impairment: serum creatinine higher than the normal reference range.
5. Allergy to band aids, adhesive dressing or medical tape.
6. Clinically significant history or presence of ECG abnormalities such as second- or third-degree atrioventricular block; evidence, or family history, of prolonged QT syndrome.
7. Sustained sitting systolic blood pressure of <90 mmHg or >140 mmHg, or diastolic blood pressure of >95 mmHg at screening or check-in of Period 1.
8. History or presence of hypersensitivity or idiosyncratic reaction to deferiprone, moxifloxacin, iron chelators, or quinolone antibiotics.
9. History or presence of:

   * agranulocytosis;
   * asthma;
   * chronic bronchitis;
   * diabetes;
   * migraine;
   * hypertension;
   * hypotension;
   * hypokalemia;
   * seizures or epilepsy;
   * anaemia.
10. History or presence of alcoholism or drug abuse within the past 2 years.
11. Used tobacco/nicotine-containing product for at least 3 months prior to the first dose of study.
12. Used Depo-Provera® or levonorgestrel implant within 90 days prior to the first dose and throughout the study.
13. Participation in another clinical trial within 28 days prior to the first dose of the study.
14. Had a clinically significant illness during the 4 weeks prior to check-in on Day -1 of Period 1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma; Caroline Fradette, PhD, Study Director — ApoPharma
Locations (1):
- Celerion, Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 17 November 2012 Last subject completed: 19 December 2012
  The study was carried out at Celerion, a research facility used for conducting clinical trials.
Groups:
- ABCD: All subjects received the same 4 treatments, separated by at least 7 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment A = single oral dose of 33 mg/kg deferiprone Treatment B = single oral dose of 50 mg/kg deferiprone Treatment C = single oral dose of placebo Treatment D = single oral dose of moxifloxacin
- BDAC: All subjects received the same 4 treatments, separated by at least 7 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment B = single oral dose of 50 mg/kg deferiprone Treatment D = single oral dose of moxifloxacin Treatment A = single oral dose of 33 mg/kg deferiprone Treatment C = single oral dose of placebo
- CADB: All subjects received the same 4 treatments, separated by at least 7 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment C = single oral dose of placebo Treatment A = single oral dose of 33 mg/kg deferiprone Treatment D = single oral dose of moxifloxacin Treatment B = single oral dose of 50 mg/kg deferiprone
- DCBA: All subjects received the same 4 treatments, separated by at least 7 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment D = single oral dose of moxifloxacin Treatment C = single oral dose of placebo Treatment B = single oral dose of 50 mg/kg deferiprone Treatment A = single oral dose of 33 mg/kg deferiprone
Period: Overall Study
Arm/Group | ABCD | BDAC | CADB | DCBA
Started | 13 | 13 | 12 | 12
Completed | 11 | 8 | 11 | 10
Not Completed | 2 | 5 | 1 | 2
Not completed — Adverse Event | 1 | 4 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Personal reason | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Fifty subjects were enrolled in order to have at least 33 subjects complete the study. The sample size calculations were based on the ICH E14 Guidance which defines a negative TQT study as one "in which the upper bound of the 95% one-sided CI for the largest time-matched mean effect of the drug on the QTc interval excludes 10 msec."
Groups:
- All Subjects: Subjects in this cross-over study all received one dose of each the following: A) a maximum therapeutic dose of 33 mg deferiprone, B) a supratherapeutic dose of 50 mg/kg deferiprone, C) placebo, and D) moxifloxacin (active control). They were randomized to receive these products in different orders: ABCD, BDAC, CADB, or DCBA. Treatments were separated by a 7-day washout period.
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Maximum Difference in Change From Baseline in ddQTcF Following a Single Dose of 33 mg/kg Deferiprone
Description: Change from baseline in QTcF interval was measured by looking at the post-dose difference in change from baseline in Fridericia's QT corrected heart rate (dQTcF) between treatment and placebo (ddQTcF) at each time interval.
  ECG recordings were obtained within a 5-minute time window at Hours -0.75, -0.5, and -0.25 (prior to dosing) and Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: Cardiodynamic Analysis Set : all randomized subjects who received at least 1 dose of study medication and who had valid Day 1 QT/QTc interval measurements (predose and at least one postdose measurement).
Measure: Least Squares Mean (Standard Deviation); unit: milliseconds
Groups:
- 33 mg/kg Deferiprone: A single dose of deferiprone 500 mg tablets at a dosage of 33 mg/kg (the maximum therapeutic level), rounded to the nearest 250 mg. Subjects additionally received deferiprone-matching placebo tablets to provide the same total number of tablets as for a 50 mg/kg dose, plus 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
- Placebo Control: A single dose of deferiprone -matching placebo tablets to provide the same total number of tablets as for a 50 mg/kg dose. Subjects additionally received 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
Arm/Group | 33 mg/kg Deferiprone | Placebo Control
Number analyzed (Participants) | 46 | 45
milliseconds | 1.4 (4.92) | -1.6 (4.72)
Statistical Analysis 1: Comparison: 33 mg/kg Deferiprone vs Placebo Control; Test type: Superiority or Other; Mean Difference (Final Values) = 3.01, 90% CI 2-sided [1.02 to 5.01]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events following therapeutic and supratherapeutic doses of deferiprone
Time Frame: From administration of the first dose until 7 days +/- 1 day following the final dose
Population: The Safety Analysis Set consisted of all subjects who received at least 1 dose of study medication and had at least 1 safety assessment.
Measure: Number; unit: participants
Groups:
- Arm A - Maximum Therapeutic Dose: A single dose of deferiprone 500 mg tablets at a dosage of 33 mg/kg (the maximum therapeutic level), rounded to the nearest 250 mg. Subjects additionally received deferiprone-matching placebo tablets to provide the same total number of tablets as for a 50 mg/kg dose, plus 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
- Treatment Arm B - Supratherapeutic Dose: A single dose of deferiprone 500 mg tablets at a dosage of 50 mg/kg (a supra-therapeutic level), rounded to the nearest 250 mg. Subjects additionally received 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
- Arm C - Placebo Control: A single dose of deferiprone-matching placebo tablets to provide the same total number of tablets as for a 50 mg/kg dose. Subjects additionally received 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
- Arm D - Positive Control: One 400 mg moxifloxacin tablet. Subjects additionally received a single dose of deferiprone-matching placebo tablets to provide the same total number of tablets as for a 50 mg/kg dose. Tablets were administered orally with approximately 240 mL of water.
Arm/Group | Arm A - Maximum Therapeutic Dose | Treatment Arm B - Supratherapeutic Dose | Arm C - Placebo Control | Arm D - Positive Control
Number analyzed (Participants) | 46 | 48 | 45 | 46
participants | 12 | 35 | 10 | 5

3. Secondary Outcome: Cmax of Deferiprone and Deferiprone 3-O Glucuronide
Description: To evaluate the Cmax of deferiprone and deferiprone 3-O-glucuronide following administration of single doses of 33 and 50 mg/kg deferiprone in healthy volunteers.
  Serial blood samples were collected prior to dosing and within 5 minutes following completion of each scheduled post-dose ECG at Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: The PK population consisted of all subjects who had taken study medication and had at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm A - Maximum Therapeutic Dose | Treatment Arm B - Supratherapeutic Dose
Number analyzed (Participants) | 46 | 48
μg/mL
  Cmax of serum deferiprone | 34.1 (8.9) | 54.4 (16.4)
  Cmax of serum deferiprone 3-O-glucuronide | 35.2 (8.5) | 51.4 (13.4)

4. Secondary Outcome: Tmax of Deferiprone and Deferiprone 3-O-glucuronide
Description: To evaluate the Tmax of deferiprone and deferiprone 3-O-glucuronide following administration of single doses of 33 and 50 mg/kg deferiprone in healthy volunteers.
  Serial blood samples were collected prior to dosing and within 5 minutes following completion of each scheduled post-dose ECG at Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: The PK population consisted of all subjects who had taken study medication and had at least 1 PK sample collected.
Measure: Median (Full Range); unit: hour
Arm/Group | Arm A - Maximum Therapeutic Dose | Treatment Arm B - Supratherapeutic Dose
Number analyzed (Participants) | 46 | 48
hour
  Tmax of serum deferiprone | 0.8185 (0.6) [0.321 to 2.13] | 0.8175 (0.9) [0.567 to 4.07]
  Tmax of serum deferiprone -O-glucuronide | 3.066 (0.7) [1.39 to 4.07] | 3.071 (0.7) [2.07 to 6.07]

5. Secondary Outcome: AUC0-infinity for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUC0-infinity was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in healthy volunteers.
  Serial blood samples were collected prior to dosing and within 5 minutes following completion of each scheduled post-dose ECG at Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: The PK population consisted of all subjects who had taken study medication and had at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: μg *hr/mL
Arm/Group | Arm A - Maximum Therapeutic Dose | Treatment Arm B - Supratherapeutic Dose
Number analyzed (Participants) | 46 | 48
μg *hr/mL
  AUC0-infinity for serum deferiprone | 95.4 (18.03) | 152.1 (22.2)
  AUC0-infinity for serum deferiprone -O-glucuronide | 205.5 (42.8) | 331.2 (74.7)

6. Secondary Outcome: T1/2 for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: T1/2 was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in healthy volunteers.
  Serial blood samples were collected prior to dosing and within 5 minutes following completion of each scheduled post-dose ECG at Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: The PK population consisted of all subjects who had taken study medication and had at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Arm A - Maximum Therapeutic Dose | Treatment Arm B - Supratherapeutic Dose
Number analyzed (Participants) | 46 | 48
hour
  T1/2 for serum deferiprone | 1.8 (0.3) | 1.8 (0.3)
  T1/2 for serum deferiprone 3-O-glucuronide | 2.5 (0.5) | 2.6 (0.2)

7. Primary Outcome: Maximum Difference in Change From Baseline in ddQTcF Following a Single Dose of 50 mg/kg Deferiprone
Description: as for outcome 1
Time Frame: 24-hour interval
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: milliseconds
Groups:
- 50 mg/kg Deferiprone: A single dose of deferiprone 500 mg tablets at a dosage of 50 mg/kg (a supra-therapeutic level), rounded to the nearest 250 mg. Subjects additionally received 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
Arm/Group | 50 mg/kg Deferiprone | Placebo Control
Number analyzed (Participants) | 48 | 45
milliseconds | 3.5 (5.28) | -1.7 (6.36)
Statistical Analysis 1: Comparison: 50 mg/kg Deferiprone vs Placebo Control; Test type: Superiority or Other; Mean Difference (Final Values) = 5.23, 90% CI 2-sided [3.26 to 7.19]

8. Primary Outcome: Maximum Postdose QT/QTc Interval
Description: The maximum post-dose QT/QTc interval for deferiprone and placebo.
  ECG recordings were obtained within a 5-minute time window at Hours -0.75, -0.5, and -0.25 (prior to dosing) and Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: The Cardiodynamic Analysis Set consisted of all randomized subjects who received at least 1 dose of study medication and who had valid Day 1 QT/QTc interval measurements (predose and at least one postdose measurement).
Measure: Number; unit: percentage of participants
Groups:
- Arm B - Supratherapeutic Dose: A single dose of deferiprone 500 mg tablets at a dosage of 50 mg/kg (a supra-therapeutic level), rounded to the nearest 250 mg. Subjects additionally received 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
- Arm C - Placebo Control: A single dose of deferiprone -matching placebo tablets to provide the same total number of tablets as for a 50 mg/kg dose. Subjects additionally received 1 moxifloxacin-matching placebo tablet. Tablets were administered orally with approximately 240 mL of water.
Arm/Group | Arm A - Maximum Therapeutic Dose | Arm B - Supratherapeutic Dose | Arm C - Placebo Control | Arm D - Positive Control
Number analyzed (Participants) | 46 | 48 | 45 | 46
percentage of participants
  QTcF ≤ 450 msec | 100 | 96 | 98 | 89
  QTcF > 450 to ≤ 480 msec | 0 | 4 | 2 | 11
  QTcF > 480 to ≤ 500 msec | 0 | 0 | 0 | 0
  QTcF > 500 msec | 0 | 0 | 0 | 0

9. Primary Outcome: Maximum Change From Baseline (dQT/dQTc)
Description: Maximum Change From Baseline (dQT/dQTc) for deferiprone and placebo.
  ECG recordings were obtained within a 5-minute time window at Hours -0.75, -0.5, and -0.25 (prior to dosing) and Hours 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 24 post-dose.
Time Frame: 24-hour interval
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Maximum Therapeutic Dose | Arm B - Supratherapeutic Dose | Arm C - Placebo Control | Arm D - Positive Control
Number analyzed (Participants) | 46 | 48 | 45 | 46
percentage of participants
  QTcF ≤ 30 msec | 100 | 100 | 100 | 96
  QTcF >30 but ≤ 60 msec | 0 | 0 | 0 | 4
  QTcF >60 msec | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Difference in Change From Baseline in ddQTcF Following a Single Dose of Moxifloxacin
Description: as for outcome 1
Time Frame: 24-hour interval
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: milliseconds
Groups:
- Positive Control: A single 400 mg tablet of moxifloxacin. The tablet was administered orally with approximately 240 mL of water.
Arm/Group | Positive Control | Placebo Control
Number analyzed (Participants) | 46 | 45
milliseconds | 14.7 (6.38) | 1.2 (6.46)
Statistical Analysis 1: Comparison: Positive Control vs Placebo Control; Test type: Superiority or Other; Median Difference (Final Values) = 13.42, 90% CI 2-sided [11.10 to 15.75]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the first dose until 7 days (± 1 day) following the last study event of Period 4 or following early withdrawal.
Groups:
- Treatment Arm A - Maximum Therapeutic Dose: Single dose of 33 mg/kg rounded to the nearest 250 mg of deferiprone tablets, deferiprone matching placebo tablets and one moxifloxacin matching placebo tablet.
  Deferiprone
  deferiprone matching placebo tablets
  moxifloxacin matching placebo tablet
- Treatment Arm B - Supratherapeutic Dose: Single dose of 50 mg/kg rounded to the nearest 250 mg of deferiprone tablets, and one moxifloxacin matching placebo tablet.
  Deferiprone
  moxifloxacin matching placebo tablet
- Treatment Arm C - Placebo Control: Single dose of deferiprone matching placebo tablets and one moxifloxacin matching placebo tablet.
  deferiprone matching placebo tablets
  moxifloxacin matching placebo tablet
- Treatment Arm D - Positive Control: Single dose of deferiprone matching placebo tablets and one 400 mg moxifloxacin tablet.
  Deferiprone
  moxifloxacin
Arm/Group | Treatment Arm A - Maximum Therapeutic Dose | Treatment Arm B - Supratherapeutic Dose | Treatment Arm C - Placebo Control | Treatment Arm D - Positive Control
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 12/46 | 35/48 | 10/45 | 5/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A - Maximum Therapeutic Dose (N=46) | Treatment Arm B - Supratherapeutic Dose (N=48) | Treatment Arm C - Placebo Control (N=45) | Treatment Arm D - Positive Control (N=46)
Palpitations (Cardiac disorders) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 19 (20) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 14 (15) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Formication (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 32 (34) | 7 (7) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All unpublished information given to the CRO by ApoPharma shall not be published or disclosed to a third party without the prior written consent of ApoPharma.

The data generated by this study are considered confidential information and the property of ApoPharma. This confidential information may be published only in collaboration with participating personnel from ApoPharma or upon ApoPharma written consent to publish the article.